CLINICAL TRIAL: NCT01573078
Title: Will The Real Psychology Of Crohn's Disease Please Stand Up?
Brief Title: Psychology of Crohn's Disease
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Robert Enns, Dr. Robert Enns, University of British Columbia
Other Study IDs: H11-02479
Record Dates: First submitted 2012-04-03; First posted 2012-04-06 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; IBS; Dissociation; Emotional processing
MeSH Terms: conditions — Crohn Disease; Dissociative Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Crohn's disease patient: Outpatients who carry a diagnosis of Crohn's disease made by a gastroenterologist.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire consisting of the following validated surveys: Rome II criteria - Scale of Body Connection (SBC), Private Body Consciousness Sub-Scale (PBCS), Body Vigilance Scale (BVS), Emotional Processing Scale (EPS25)

SUMMARY:
The purpose of this study is to determine whether emotional processing and somatic dissociation influence IBS-like symptoms in Crohn's Disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Age of 19 or greater
* Outpatient with diagnosis of Crohn's disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Crohn's Disease Patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2015-01-28 (Actual); Study Completion 2015-01-28 (Actual)

PRIMARY OUTCOMES:
presence of functional gastrointestinal disorder | within previous 6 months

SECONDARY OUTCOMES:
difference in ability to process emotions | within previous 6 months
difference in body awareness and degree of bodily-dissociation | within previous 6 months
difference in sensitivity to internal bodily sensations | within previous 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Enns, MD, Principal Investigator — University of British Columbia
Locations (1):
- Pacific Gastroenterology Associates, Vancouver, British Columbia, Canada